CLINICAL TRIAL: NCT03616067
Title: Evaluation of the Long-term Efficacy of the Injection of Botulinum Toxin A Into the Salivary Glands Versus Scopolamine Patches in the Treatment of Drooling in Children Over 4 Years Old With Cerebral Palsy.
Brief Title: Evaluation of the Efficacy of the Injection of Botulinum Toxin A vs Scopolamine Patches in the Treatment of Drooling in Children With Cerebral Palsy
Acronym: TOXSIALO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Steering Committee decided on 22/09/2025 to end the project, due to persistent issues: enrolment suspended because of supply shortages and the arrival of alternative treatments, as well as the end of a key supply agreement.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0235
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox® injection arm (Experimental): Botox® injection in salivary glands will be performed one month after inclusion. It will be performed with one injection point per gland (parotids and submandibulars).
  Interventions: Drug: Botox® injection
- Scopoderm® patches arm (Active Comparator): Scopoderm® patches will be initiated one month after inclusion. The patches will be renewed every 3 days, alternating behind each ear
  Interventions: Drug: Scopoderm® patches arm

INTERVENTIONS:
Drug: Botox® injection — Botox® injection in salivary glands will be performed one month after inclusion. It will be performed with one injection point per gland (parotids and submandibulars)
  Arms: Botox® injection arm
Drug: Scopoderm® patches arm — Scopoderm® patches will be initiated one month after inclusion. The patches will be renewed every 3 days, alternating behind each ear.
  Arms: Scopoderm® patches arm

SUMMARY:
Cerebral palsy is the first cause of motor disability in developed countries. It is associated with altered motor function but also with mental, sensorial and behavior deficiencies. Drooling frequently occurs in children with cerebral palsy (37 to 58%). It causes multiple medical and social complications which can all increase disability and reduce quality of life for the patients and their family. Drooling treatments are various and includes orofacial rehabilitations, anticholinergic medications, botulinum toxin A and B salivary gland injections. Surgeries could also be used, but their benefits are often outweighed by the risk.

* Orofacial rehabilitation is firstly recommended, even if few studies evaluated its efficacy.
* Medication by Scopoderm®, a cutaneous anticholinergic drug, is frequently used in spite of frequent side effects and a lack of evidence regarding efficacy.
* Botulinum toxin salivary gland injections (Botox®) were shown to be effective in reducing the severity of drooling consequences for the patient quality of life up to 12 months after the injections (Reid 2008).

A recent survey carried showed that treatment by Botox® injection would be preferred by professional to Scopoderm® patch, because of better tolerance and efficacy, even if Scopoderm® remained more used by professionals (Chaleat-Valayer 2016). However, a Cochrane review (Walshe 2012) concluded that there is 1) no strong consensus regarding assessment or the timing of all treatments 2) not enough efficacy studies with high level of evidence, 3) mostly efficacy studies vs placebo or no intervention 4) a lack of long term treatment assessment 5) a lack of studies on the patient quality of life.

Our study will be a comparative randomized clinical trial with an active control arm. The hypothesis is that therapeutic treatment of drooling in children with cerebral palsy consisting of a standardized rehabilitation treatment associated with a botulinum toxin A injection (Botox®) in the salivary glands is more effective than the same rehabilitation treatment associated with a treatment by scopolamine patches (Scopoderm®).

The main outcome will be assessed 15 months after initiation of treatment to evaluate long-term effectiveness. Patients from both arms of the trial will received rehabilitation, in order to compare treatment efficacy as it is done in real conditions of treatment. The efficacy of the treatment will be assessed on the impact of the drooling perceived by the patients and their family rather than on the measure of salivary production, as recommended (Walshe 2012).

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 to 18 years old,
* Cerebral palsy with pathological drooling,
* Significant impact of drooling on the children (DIS score ≥40),
* Affiliated or beneficiary of a social security scheme,
* At least one of the parents understanding and speaking French,
* Written consent form signed by both parents

Exclusion Criteria:

* Previous history of surgery for drooling,
* Injection of botulinum toxin (all locations) in the 3 months prior to the inclusion,
* Treatment by scopolamine patch (Scopoderm®) or other anticholinergic (Artane®, etc.) in the month prior to inclusion,
* Contraindication to the anesthetic or sedation,
* Contraindication to one of the treatments studied (glaucoma, myastenia),
* Swallowing disorder (to saliva) or absence of spontaneous swallowing reflex not investigated by nasoscopy
* On-going or programmed orthodontic treatment over the study period.
* Untreated oro-mandibular dystonia (isolated lingual dystonia accepted)
* Untreated bruxism
* Untreated clinical gastro esophageal reflux
* Untreated dental inflammatory condition (dental caries, gingivitis…)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Drooling Impact Scale (DIS scale) | after 15 months of treatment
  The DIS scale is a questionnaire of 10 questions with a score of 100 points which will be completed by the patient's entourage (family and/or caregivers). This scale has a good validity and sensitivity to changes in the context of the evaluation of the drooling in children with CP, with a score difference of 10 points considered as clinical significant.

SECONDARY OUTCOMES:
DIS scale | at 1, 3, 6, 9 and 12 months of treatment
  The DIS scale is a questionnaire of 10 questions with a score of 100 points which will be completed by the patient's entourage (family and/or caregivers). This scale has a good validity and sensitivity to changes in the context of the evaluation of the drooling in children with CP, with a score difference of 10 points considered as clinical significant
Drooling severity | at 1, 3, 6, 9, 12 and 15 months of treatment
  average number of bibs used per day per patient
Clinical complications of the drooling | at 1, 3, 6, 9, 12 and 15 months of treatment
  The number of hospitalizations for pulmonary infections and the average number of prescriptions for antibiotic treatment linked to bronchial secondary infection.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine TOUZET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (11):
- France (11):
  - CHU d'Angers, Angers
  - CHU-Bordeaux, Bordeaux
  - Hôpital Femme Mère Enfant - HCL, Bron
  - CHU- Estaing, Clermont-Ferrand
  - CHU-Grenoble, Grenoble
  - Centre Médico-Chirurgical de Réadaptation des Massues, Lyon
  - AP-HM, Marseille
  - APFESEAN Nantes, Nantes
  - CHU-Nimes, Nîmes
  - Centre médico- infantile, Romagnat
  - Hôpitaux de Saint-Maurice, Saint-Maurice

IPD SHARING:
Plan to Share IPD: No